CLINICAL TRIAL: NCT02151409
Title: A Randomised, Double-blind, Placebo-controlled, Single-dose, Dose-escalation Trial of Anti-C5aR Antibody (NNC 0151-0000-0000) Administered by i.v. Infusion or s.c. Injection in Healthy Subjects.
Brief Title: Dose-escalation Trial of Anti-C5aR Antibody in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN8209-1940; 2008-000731-18 (EudraCT Number)
Record Dates: First submitted 2014-05-28; First posted 2014-05-30 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Inflammation; Systemic Lupus Erythematosus; Rheumatoid Arthritis; Healthy
MeSH Terms: conditions — Inflammation; Lupus Erythematosus, Systemic; Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- NNC 0151-0000-0000 i.v. (Experimental): Dose escalation trial
  Interventions: Drug: NNC 0151-0000-0000
- NNC 0151-0000-0000 s.c. (Experimental): Dose escalation trial
  Interventions: Drug: NNC 0151-0000-0000
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: NNC 0151-0000-0000 — A single dose (SD), administrated i.v. (intravenous) at 8 dose levels.
  Arms: NNC 0151-0000-0000 i.v.
Drug: NNC 0151-0000-0000 — A single dose (SD), administrated s.c. (subcutaneously) at 7 dose levels
  Arms: NNC 0151-0000-0000 s.c.
Drug: placebo — A single dose (SD), administrated i.v. (intravenous) or s.c. (subcutaneously).
  Arms: Placebo

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to develop a complement system targeted monoclonal antibody (mAb) to be used in treatment of subjects with chronic autoimmune diseases.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities (Trial-related activities are any procedure that would not have been performed during normal management of the subject)
* Body weight (BW) below or equal to 110.0 kg
* Body Mass Index (BMI) 20.0 - 27.0 kg/m^2, both inclusive
* Good state of health: evidenced by medical history, physical examination and results of laboratory examinations

Exclusion Criteria:

* History of known or suspected cardiovascular diseases including: supine systolic blood pressure (BP) above or equal to 140 mmHg or below 90 mm Hg, diastolic BP above oe equal to 90 mm Hg or below 40 mm Hg, heart rate (HR) in supine position above 100 beats/minute or below 45 beats/minute
* Hepatic insufficiency: Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) above Upper Limit of Normal (ULN) (retesting is permitted within one week if first test is elevated but below 1.5 fold ULN)
* Renal insufficiency: Serum creatinine above ULN
* Positive for humane immunodeficiency virus (HIV) (by test)
* Positive for hepatitis B (HBV) or hepatitis C (HCV) (by test)

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2008-06; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Adverse events (AEs) | Week 0-10

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Groningen, Netherlands

REFERENCES:
- [Result] The first-in-human trial of the humanised monoclonal antibody NNC 0151-0000-0000 blocking the C5a receptor (C5aR). EULAR (European League Against Rheumatism) 2009; Country: Denmark City: Copenhagen
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com